CLINICAL TRIAL: NCT06152133
Title: Effects of a Telerehabilitation Program of Central Stability Exercises to Improve Balance and Gait in Hereditary Ataxia. A Randomized Controlled Pilot Study.
Brief Title: Telerehabilitation, Core Stability Exercises and Hereditary Ataxia (TRCore-ataxia)
Acronym: TRCore-ataxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat de Lleida (Other)
Collaborators: Universitat Internacional de Catalunya (Other); Hospital Clinic of Barcelona (Other); Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Maria Masbernat-Almenara, Principal Investigator, Universitat de Lleida
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Hereditary Ataxia; Spinocerebellar Degenerations; Cerebellar Ataxia
Keywords: Spinocerebellar Degenerations; Telerehabilitation; Exercise
MeSH Terms: conditions — Spinocerebellar Degenerations; Cerebellar Ataxia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Pilot
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telerehabilitation Core stability exercises group (Experimental)
  Interventions: Other: Therapeutic core stability exercises
- Core stability exercises group (Active Comparator)
  Interventions: Other: Therapeutic core stability exercises

INTERVENTIONS:
Other: Therapeutic core stability exercises — exercises focused on trunk muscle strengthening, proprioception, selective movements of the trunk and pelvis muscle, and coordination, and will be carried out in supine, sitting on a stable surface and sitting on an unstable surface (ball). The exercise involves changes in the position of the body with or without resistance, aiming to improve strength, endurance, proprioception and coordination. Training is determined by the patient's ability to undertake easy exercises and progress to more challenging exercises.
  Other Names: trunk exercises

SUMMARY:
Hereditary ataxias (HA) are a heterogeneous group of degenerative diseases of the cerebellum, brain stem and spinal cord. People who suffer from AH, among other symptoms, present deficiencies in the stability of the trunk, which leads to an alteration in postural control, with a strongly influential factor in the loss of balance and gait disorders. Improving the functionality of these physical aspects can help reduce the rate of falls, increase autonomy and quality of life for people with HA.

Evidence suggests that rehabilitation strategies based on core stability exercises (CSE) are effective in improving balance and postural control in several neurological diseases, such as stroke. However, there is little evidence with people with HA. In a previous study carried out by researchers of this project, in which an EEC exercise program was piloted at home, low adherence to treatment was perceived due to the little follow-up that was given to the participants. Therefore, including telerehabilitation in these programs would increase follow-up and could influence adherence.

ELIGIBILITY:
Inclusion Criteria:

* Suffer from degenerative HA at any stage of the disease (Spinocerebellar ataxia, Friedreich's ataxia, sporadic idiopathic cerebellar ataxia and neurodegenerative diseases where ataxia is the dominant symptom).
* Adults over 18 years of age.
* Be able to use a computer or mobile phone (It will be evaluated using the DILE scale)
* Have an internet connection.

Exclusion Criteria:

* Suffer from other neurological diseases and inability to follow simple instructions. -
* Suffering from a musculoskeletal injury that prevents you from performing the exercises.
* Being unable to maintain standing for more than 10 seconds without support (assessed with item 2 on the SARA scale).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Rate of dynamic sitting balance and trunk coordination | T0: Baseline, T1: 7 weeks and T0: follow up 7 weeks
  panish-version of Trunk Impairment Scale 2.0. Each item will be performed three times and the highest score counts. Otherwise, no practice session allowed. The patient can be corrected between attempts. The tests are verbally explained to the patient and can be demonstrated if needed. There are two subscales: dynamic sitting balance and coordination. The first have 10 items and second 6. The highest possible total score is consequently 16 points, which indicates a good dynamic sitting balance and correct trunk control and sitting coordination. If the patient cannot maintain a sitting position for 10 seconds without back and arm support, with hands on thighs, feet in contact with the ground and knees bent at 90° (starting position), the total score for the scale is 0 points.
Static sitting balance and Standing balance | T0: Baseline, T1: 7 weeks and T0: follow up 7 weeks
  Static sitting balance will be recorded with the sitting section of SARA, standing balance will be recorded with the standing section of SARA as well, as well as walking.
Walking Speed | T0: Baseline, T1: 7 weeks and T0: follow up 7 weeks
  The walking speed will be determined with the 4 meter walking test.

SECONDARY OUTCOMES:
ADLs | T0: Baseline, T1: 7 weeks and T0: follow up 7 weeks
  ADLs will be assessed with the Activities-specific Balance Confidence (ABC)
Lower extremity strength | T0: Baseline, T1: 7 weeks and T0: follow up 7 weeks
  Lower extremity strength will be assessed with the 30 s Sit-to-stand test.
Adherence to treatment | T1: 7 weeks and T0: follow up 7 weeks
  Adherence to treatment will be asses with the Exercise Adherence Rating Scale (EARS) (Newman-Beinart 2017).
Risk of falls | T0: Baseline, T1: 7 weeks and T0: follow up 7 weeks
  The risk of falls with the Timed Up and GO scale
Severity of ataxia | T0: Baseline, T1: 7 weeks and T0: follow up 7 weeks
  The severity of ataxia will be evaluated with the SARA scale
Treatment compliance | T1: 7 weeks and T0: follow up 7 weeks
  treatment compliance measured as the rate of sessions performed/prescribed (Capecci 2023), we will obtain the % compliance for each participant with the calculation Total number of minutes performed by the patient / Total number of minutes that should have been done (1400 minutes) x 100. Or with the calculation Total number of exercises per session performed by the patient / Total number of exercises that should have been done (23 per session) x 100
Program satisfaction | T1: 7 weeks
  A questionnaire will be administered to participants to evaluate both their experience and satisfaction with the program, as well as its adverse effects.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Lleida, Lleida, Lleida, Spain

IPD SHARING:
Plan to Share IPD: Yes